CLINICAL TRIAL: NCT07292558
Title: Achieving Health in Emerging Adults With Diabetes (AHEAD) Study
Brief Title: Achieving Health in Emerging Adults With Diabetes (AHEAD) Program: A Clinical Trial Designed to Understand if Participation in a Clinical Program Developed Specifically to Support Emerging Adults With Type 1 Diabetes Leads to Improved Diabetes Outcomes.
Acronym: AHEAD Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Breakthrough T1D (Other); Seattle Children's Hospital (Other); University of Washington (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Faisal Malik, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H25-03574; 4-SRA-2024-1580-M-B (Other Grant/Funding Number: Breakthrough T1D)
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1 Diabetes
Keywords: Adolescent; Young adult; Emerging adult; Patient transfer; Health care transition; Transition readiness; Diabetes self-management; Diabetes distress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AHEAD Program (Experimental): AHEAD participants will receive support from a team of diabetes providers with expertise in supporting older adolescents and young adults who will work to build autonomy and competence needed to manage diabetes independently.
  Interventions: Behavioral: AHEAD Program
- Usual Care (No Intervention): Usual Care participants will receive diabetes care as currently being provided by their primary medical team.

INTERVENTIONS:
Behavioral: AHEAD Program — Participants will complete self-assessments around health care transition readiness and mental health prior to an AHEAD clinic visit. Emerging adults will then received tailored clinical support based on their self-assessments and work to build their autonomy and competence to manage their diabetes and health care independently with the support of their AHEAD providers.
  Arms: AHEAD Program

SUMMARY:
The goal of this study is to determine whether the Achieving Health in Emerging Adults with Diabetes (AHEAD) Program helps emerging adults with type 1 diabetes improve their blood glucose management during the transition from pediatric to adult care.

Participants will be randomized to receive Usual Care or the AHEAD Program, which provides tailored support to emerging adults to build autonomy and competence to facilitate independent diabetes management. Researchers will compare changes in glycemia and participant-reported outcomes between groups.

DETAILED DESCRIPTION:
Many emerging adults with type 1 diabetes find it difficult to maintain their blood glucose levels within the recommended range most of the time. This can increase their risk for serious short- and long-term diabetes-related health problems. Managing diabetes becomes especially difficult during the transition from pediatric care to adult care when emerging adults are expected to manage their condition on their own.

The Achieving Health in Emerging Adults with Diabetes (AHEAD) Program was developed to support emerging adults with their transition to independence. It focuses on helping them build autonomy and competence needed to manage their diabetes independently. The program is based on self-determination theory and best practices for supporting successful health care transition to adult care.

In this study, 306 emerging adults will be randomly assigned to either the AHEAD Program or Usual Care arms. Participants will have 6 clinic visits and complete surveys prior to their clinic visits. AHEAD participants will receive support from a team of diabetes providers who have expertise in supporting emerging adults living with diabetes every three months. Usual Care participants will continue to receive the diabetes care as they do currently every three months.

Researchers will evaluate changes in glycemia and participant-reported outcomes (e.g., diabetes distress, transition readiness). The study will also assess the cost and cost-effectiveness of AHEAD, as well as factors related to its implementation.

ELIGIBILITY:
Inclusion Criteria:

1. 16-19 years of age
2. Have had type 1 diabetes ≥ 12 months
3. Had a recent HbA1c ≥7.0%
4. Currently receive outpatient diabetes care at a Seattle Children's Hospital Diabetes Clinic located in Bellevue, Everett, Federal Way, or Seattle
5. Are able to complete written surveys
6. Will be able to receive clinical care in WA State for the next 2 years

Exclusion Criteria:

1. Have had a pilot program AHEAD clinic visit
2. Most recent Usual Care diabetes visit was with a current AHEAD provider

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  HbA1c laboratory measurement.

SECONDARY OUTCOMES:
Time In Ranges | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Continuous glucose monitor sensor glucose measurements that are in range (70-180 mg/dL), above range (>180 mg/dL), and below range (<70 mg/dL).
Diabetes Distress | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Diabetes distress will be assessed with the Problem Areas in Diabetes Scale -- Teen Version. Higher scores indicate higher diabetes distress (score: 14-84).
Diabetes-Specific Health Care Transition Readiness | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Diabetes-specific health care transition readiness will be assessed with the Readiness Assessment of Emerging Adults with Type 1 Diabetes tool. Higher scores (mean topic area score: 1-5) indicate higher diabetes-specific transition readiness.
General Health Care Transition Readiness | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  General health care transition readiness will be assessed with the Transition Readiness Assessment Questionnaire. Higher scores (mean topic area score: 1-5) indicate higher transition readiness.
Diabetes Family Conflict | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Diabetes family conflict will be assessed with the Diabetes Family Conflict Scale. Higher scores indicate higher diabetes family conflict (score: 19-57).
Relatedness | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Relatedness will be measured using the Health Care Climate Questionnaire. Higher scores indicate more supportive health care practitioner(s) (score: 15-105).
Autonomy Treatment Self-Regulation Questionnaire | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Autonomy will be measured using the Treatment Self-Regulation Questionnaire. Higher scores indicate higher autonomy (score: 15-105).
Disordered eating | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Disordered eating will be measured using the Disordered Eating Problem Survey - Revised. Higher scores indicate increase disordered eating behaviors (score: 0-80).
Depression | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Depression will be measured using the Patient Health Questionnaire-9. Higher scores indicate higher depression severity (score: 0-27).
Generalized Anxiety | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Anxiety will be measured using the Generalized Anxiety Disorder-7 questionnaire. Higher scores indicate higher severity of anxiety (score: 0-21).
Social needs | From enrollment (baseline clinic visit: 0 months) to the end of intervention period (6th clinic visit: 15-24 months).
  Social needs will be measured using the social needs questionnaire. Endorsement of financial insecurity, food insecurity, transportation challenges, and housing insecurity, will indicate higher social need(s) (score: N/A).

CONTACTS AND LOCATIONS:
Overall Officials: Faisal S Malik, MD, MSc, Principal Investigator — University of British Columbia
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be stored in a publicly available repository (OpenScience Framework: https://osf.io/). To address privacy and confidentiality concerns, sharing of data generated will be limited to de-identified data at the aggregate level.
Supporting Information: SAP
Time Frame: Data requests can be submitted at the end of the funding period and the data will be made accessible for up to 10 years.
Access Criteria: Access, distribution, and reuse of the data will require approval from study investigators.